CLINICAL TRIAL: NCT07007130
Title: Effect of Intraperitoneal Insulin Administration After Laparoscopy in Insulin-Resistant Patients on Prevention of Postoperative Adhesion Recurrence: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Asisstant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Dr Sayed Elakhras study
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Prevention of Postoperative Adhesions
MeSH Terms: interventions — insulin, neutral; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator)
  Interventions: Drug: Actrapid insulin
- Control group (Sham Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Actrapid insulin — 0.1 IU/kg of short-acting human insulin diluted in 100 mL of normal saline, instilled intraperitoneally before closure
  Arms: Intervention group
Drug: Normal saline — 100 mL normal saline intraperitoneally
  Arms: Control group

SUMMARY:
Adhesion formation following laparoscopic pelvic surgery remains a significant cause of chronic pelvic pain, infertility, and surgical complications. Patients with insulin resistance (IR) may have heightened inflammatory responses and impaired tissue healing, contributing to a higher risk of adhesion formation. Intraperitoneal administration of insulin has shown promising results in animal models by modulating inflammatory mediators and enhancing fibrinolysis. This trial aims to evaluate the efficacy and safety of intraperitoneal insulin instillation at the end of laparoscopy in women with insulin resistance.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, double-blind clinical trial designed to evaluate the efficacy of intraperitoneal insulin administration at the end of laparoscopic surgery in women with insulin resistance, aiming to reduce postoperative adhesion formation. The study will be conducted at a dr saed hospital and will enroll 100 female patients diagnosed with insulin resistance undergoing laparoscopy for infertility or chronic pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years
* Diagnosed insulin resistance (e.g., HOMA-IR >2.5 or fasting insulin >15 uIU/mL)
* Indicated for laparoscopy for infertility or pelvic pain
* BMI 20-35 kg/m²
* Able and willing to give informed consent

Exclusion Criteria:

* Diabetes mellitus requiring pharmacologic treatment
* History of peritonitis or major abdominal surgery in the past 6 months
* Known allergy or sensitivity to insulin
* Chronic steroid or immunosuppressive use
* Pregnancy or lactation
* Participation in another clinical trial within the last 3 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Adhesion scoring at second-look laparoscopy | 4-6 weeks postoperatively
  Adhesion scoring at second-look laparoscopy (4-6 weeks postoperative)

SECONDARY OUTCOMES:
Postoperative pain scores | Immediately after operation
Hypoglycemic events | 2 hours after the operation
Hypoglycemic events | 4 hours after the operation
Fertility rates | At 6 months